CLINICAL TRIAL: NCT00098605
Title: A Phase 2 Study of GW572016 for Brain Metastases in Patients With HER2-Positive Breast Cancer
Brief Title: Lapatinib in Treating Brain Metastases in Patients With Stage IV Breast Cancer and Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02934; DFCI 04-199
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Central Nervous System Metastases; HER2-positive Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer; Tumors Metastatic to Brain
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Brain Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

ARMS (1):
- Treatment (lapatinib ditosylate) (Experimental): Patients receive oral lapatinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Drug: lapatinib ditosylate — Given orally
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Other: laboratory biomarker analysis — Correlative studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for their growth. This phase II trial is studying how well lapatinib works in treating brain metastases in patients with stage IV breast cancer and brain metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate in the central nervous system (CNS) (complete plus partial responses), as assessed by standard MRI, to oral GW572016 among patients with progressive brain metastases from HER2-positive breast cancer.

SECONDARY OBJECTIVES:

I. To evaluate the site of first failure (CNS, extra-CNS, both, or death) and overall survival of patients treated with GW572016 for brain metastases.

II. To evaluate the overall objective response rate (complete plus partial response) and time to first progression at any site.

III. To assess quality of life (QOL), neurologic QOL, and cause of death in patients treated with GW572016 for brain metastases.

IV. To determine the qualitative and quantitative toxicities associated with oral GW572016, given at a dose of 750 mg orally, twice daily.

V. To evaluate the sensitivity of PET with dedicated brain sequences to detect brain metastases from breast cancer.

VI. To explore the relationship between decline in PET uptake at 1 week and decline in PET uptake at 8 weeks.

VII. To characterize the vessel patterns seen on MRI at baseline, 8 weeks, and 16 weeks of treatment with GW572016.

VIII. To describe changes in serum HER2 ECD over time. IX. To describe the baseline EGFR, HER2, IGF-IR, and degree of HER2 gene amplification in primary tumor blocks.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral lapatinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and at 8 weeks.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 0.5-1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed invasive breast cancer, with stage IV disease
* HER2 overexpressing breast cancer, defined as 3+ staining by immunohistochemistry (IHC), or 2+ staining by IHC in conjunction with HER2 gene amplification by fluorescent in situ hybridization (FISH), or HER2 gene amplification by FISH alone (in patients whose tumor blocks were not assessed by IHC); patients with tumors that are 2+ by IHC but negative by FISH assay are ineligible
* At least one measurable lesion in the CNS, defined as any lesion >= 10 mm in longest dimension on T1-weighted, gadolinium-enhanced MRI
* One of the following:

  * Cohort 1: Prior treatment of CNS metastases with whole brain radiotherapy (WBRT) and/or stereotactic radiosurgery (SRS), OR;
  * Cohort 2: Asymptomatic CNS metastases discovered on a screening radiological study without prior WBRT or SRS
* Disease progression in the CNS, as assessed by at least one of the following:

  * New neurological signs or symptoms
  * New lesions in the CNS on an imaging study
  * Progressive lesions on an imaging study
  * Note: patients with progressive lesions are not required to meet Response Evaluation Criteria in Solid Tumors (RECIST) criteria for progression in order to be eligible for this study
* Prior treatment with trastuzumab, either alone or in combination with chemotherapy is required; trastuzumab will be discontinued at least 2 weeks prior to enrollment on study; note: patients who have documented CNS-only metastases are not required to have had prior treatment with trastuzumab; in this situation, the absence of extra-CNS disease must be documented with a physical examination, CT scan of the chest, abdomen, and pelvis, and bone scan
* At least 2 weeks since prior radiotherapy, last chemotherapy, immunotherapy, biologic therapy, or hormonal therapy for cancer, and sufficiently recovered or stabilized from side effects associated with prior therapy; concurrent treatment with bisphosphonates is permitted
* At least 3 weeks since major surgical procedures
* At least 2 weeks since last dose of trastuzumab
* Life expectancy >= 12 weeks
* ECOG performance status 0-2 (Karnofsky >= 60%)
* Hemoglobin >= 9 g/dL (after transfusion if needed)
* Platelets >= 50 x 10^9/L
* Albumin >= 2.5 g/dL
* Serum bilirubin =< 1.5 x ULN unless due to Gilbert's syndrome
* AST and ALT =< 5 x ULN
* Serum creatinine =< 1.5 mg/dL or calculated creatinine clearance >= 25 mL/min (calculated by the Cockcroft and Gault method)
* Cardiac ejection fraction within institutional normal limits, as assessed by echocardiogram or MUGA scan
* Women of childbearing potential are eligible for this study provided they agree to one of the following:

  * Complete abstinence from intercourse from 2 weeks prior to administration of the first dose of GW572016 until 28 days after the final dose of GW572016; or
  * Consistent and correct use of one of the following acceptable methods of birth control:
  * Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; or
  * Implants of levonorgestrel
  * Injectable progestogen
  * Any intrauterine device (IUD) with a documented failure rate of less than 1% per year; or
  * Oral contraceptives (either combined or progestogen only)
  * Barrier methods including diaphragm or condom with a spermicide Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Able to swallow and retain oral medications
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or who have unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment
* Patients may not be receiving any other investigational agents
* Patients may not be receiving concurrent chemotherapy, radiation therapy, immunotherapy, biologic therapy (including an ErbB1 and/or ErbB2 inhibitor), or hormonal therapy for treatment of their cancer; concurrent treatment with bisphosphonates is allowed
* Patients with leptomeningeal carcinomatosis as the only site of CNS involvement will be excluded from this clinical trial, because disease is not measurable, and standard treatment options may differ
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GW572016
* Concurrent treatment with medications that are either inducers or inhibitors of CYP3A4 is prohibited; some common examples are phenytoin, carbamazepine, and phenobarbital; if a patient requires an anticonvulsant, valproic acid or levetiracetam (Keppra) may be substituted, under the direction of his/her treating physician and/or neurologist
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel; subjects with active ulcerative colitis are also excluded
* History of immediate or delayed hypersensitivity reaction to gadolinium contrast agents, or other contraindication to gadolinium contrast
* Other known contraindication to MRI, such as a cardiac pacemaker, implanted cardiac defibrillator, brain aneurysm clips, cochlear implant, ocular foreign body, or shrapnel
* Concurrent disease or condition that would make the subject inappropriate for study participation, or any serious medical or psychiatric disorder that would interfere with the subject's safety
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Pre-existing severe cerebral vascular disease, such as stroke involving a major vessel, CNS vasculitis, or malignant hypertension
* Active cardiac disease, defined as:

  * History of uncontrolled or symptomatic angina
  * History of arrhythmias requiring medications, or clinically significant, with the exception of asymptomatic atrial fibrillation requiring anticoagulation
  * Myocardial infarction < 6 months from study entry
  * Uncontrolled or symptomatic congestive heart failure
  * Ejection fraction below the institutional normal limit
  * Any other cardiac condition, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
* Active or uncontrolled infection
* History of other malignancy, except for curatively treated basal cell carcinoma or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix; subjects with other malignancies who have been disease-free for at least 5 years are eligible
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with GW572016

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-10; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate defined as the percentage of patients with a complete response (CR) or partial response (PR) in the CNS | Up to 5 years
  A 95% confidence interval (CI) for percent of patients with CNS response will be calculated if the study does not terminate accrual early. The method of Atkinson and Brown will be used to calculate the CI conditional on the sequential design.

SECONDARY OUTCOMES:
Objective response in non-CNS sites | Up to 5 years
  A 95% CI for percent of patients with CNS response will be calculated if the study does not terminate accrual early. The method of Atkinson and Brown will be used to calculate the CI conditional on the sequential design.
Site of first progression | At the time of disease progression
Time to progression (TTP) | From study entry to the first documented evidence of disease progression, assessed up to 5 years
  The time to progression will be summarized using a Kaplan-Meier survival curve.
Overall survival | From study entry until death due to any cause, assessed up to 5 years
  Overall survival for each cohort will be summarized using a Kaplan-Meier survival curve.
Quality of life assessed using the European Organization for the Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire Core Cancer Module (QLQ-C30) and EORTC Brain Cancer Module (BCM-20) | Baseline
  Changes from baseline will be summarized for the total score and subscale scores. Responses will be scored and reported according to published methods. The baseline and change scores will be characterized descriptively.
Quality of life assessed using the EORTC QLQ-C30 and EORTC BCM-20 | Week 8
  Changes from baseline will be summarized for the total score and subscale scores. Responses will be scored and reported according to published methods. The baseline and change scores will be characterized descriptively.
Cause of death classified as being due to systemic disease progression, primarily due to CNS disease progression, primarily due to treatment-related toxicity, or unrelated to the subject's breast cancer diagnosis | Up to 5 years
  The proportion of patients who fall into each category will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Winer, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States